CLINICAL TRIAL: NCT03712748
Title: Imaginal Exposure I Online Study
Brief Title: Online Imaginal Exposure
Acronym: Online IE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Cheri Levinson, Director, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#:16.0771
Record Dates: First submitted 2018-06-20; First posted 2018-10-19 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Eating Disorder; Exposure; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder | interventions — Implosive Therapy

STUDY DESIGN:
Intervention Model Description: All participants will complete the same arm, which is four sessions of imaginal exposure across a one month time period. Each session is separated by 1 week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginal Exposure Session (Experimental)
  Interventions: Behavioral: Imaginal Exposure therapy

INTERVENTIONS:
Behavioral: Imaginal Exposure therapy — All participants will complete the same arm, which is four sessions of imaginal exposure across a one month time period. Each session is separated by 1 week.
  Other Names: Exposure Therapy

SUMMARY:
This study evaluates if imaginal exposure therapy can decrease symptoms of eating disorders and anxiety, and test an online format of IE to maximize its ability to reach as many individuals with eating disorders as possible. All participants will complete four imaginal exposure sessions and will complete questionnaires prior to receiving this treatment, as well as complete follow up questionnaires at 1-month, 6-month, and 12-month.

DETAILED DESCRIPTION:
Eating disorders (EDs) are tenacious mental disorders that are difficult to treat. EDs are often accompanied by anxiety disorders, which exacerbate the problem. Better ED treatments are imperative, and it is likely that targeting comorbid conditions, such as anxiety, will facilitate ED treatments.

Imaginal exposure is used in anxiety disorders to face fears that are not accessible or practical to address via in-vivo exposures. For example, a patient with PTSD cannot re-experience her trauma in real life, but she can imagine the past trauma and experience the subsequent anxiety. For patients with AN, catastrophic outcomes such as abandonment or immediate fatness are similarly impossible to recreate as in-vivo exposures. Patients cannot become fat solely for the purpose of the exposure, but they can imagine what it would be like to become fat. The investigators are unaware of any literature using imaginal exposure therapy to induce fears of fatness and conducted a case study to test whether imaginal exposure could, firstly, induce fears of fatness and then promote reduction in anxiety and eating disorder symptoms. In this case study, the investigators found that imaginal exposure therapy was effective at reducing anxiety and eating disorder behaviors. Imaginal exposure therapy (IE) has been shown to be an extremely effective treatment for Post-Traumatic Stress Disorder. IE has also been shown to be effective for the treatment of eating disorders using case studies. However, IE has not been systematically applied to the eating disorders. The purpose of this study is to test if 1) imaginal exposure therapy can decrease symptoms of eating disorders and anxiety, and 2) test an online format of IE to maximize its ability to reach as many individuals with eating disorders as possible.

ELIGIBILITY:
Inclusion Criteria:

* At least 14 years of age (no age limit)
* Currently meet criteria for an eating disorder (using the eating disorder diagnostic scale), OR have met criteria for an eating disorder in the last year, OR endorse significant eating disorder fears
* At least one significant eating disorder related fear.

Exclusion Criteria:

* Under 14 years of age
* Do not meet eating disorder related criteria
* Do not meet criteria for mania, psychosis, or suicidal ideation will be excluded.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms are assessed by the Eating Disorder Examination Questionnaire | Up to 12 Months
  The Eating Disorder Examination Questionnaire (EDEQ), a self-reported measure, is assessed at multiple time points throughout the duration of the study and is used to examine the attitudes and behaviors in individuals with eating disorder symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Anxiety Treatment Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Rapp J, Riley EN. Addressing the fear of fat: extending imaginal exposure therapy for anxiety disorders to anorexia nervosa. Eat Weight Disord. 2014 Dec;19(4):521-4. doi: 10.1007/s40519-014-0115-6. Epub 2014 Apr 2. No abstract available. PMID 24691784
- [Background] Steinglass JE, Sysko R, Glasofer D, Albano AM, Simpson HB, Walsh BT. Rationale for the application of exposure and response prevention to the treatment of anorexia nervosa. Int J Eat Disord. 2011 Mar;44(2):134-41. doi: 10.1002/eat.20784. PMID 20127936
- [Background] Steinglass JE, Albano AM, Simpson HB, Wang Y, Zou J, Attia E, Walsh BT. Confronting fear using exposure and response prevention for anorexia nervosa: A randomized controlled pilot study. Int J Eat Disord. 2014 Mar;47(2):174-80. doi: 10.1002/eat.22214. Epub 2013 Nov 8. PMID 24488838
- [Derived] Levinson CA, Christian C, Ram SS, Vanzhula I, Brosof LC, Michelson LP, Williams BM. Eating disorder symptoms and core eating disorder fears decrease during online imaginal exposure therapy for eating disorders. J Affect Disord. 2020 Nov 1;276:585-591. doi: 10.1016/j.jad.2020.07.075. Epub 2020 Jul 21. PMID 32794449